CLINICAL TRIAL: NCT03032757
Title: Defining the Role of Lysosomal Movement in Age-associated Anabolic Resistance in Human Skeletal Muscle
Brief Title: Lysosomal Movement and Anabolic Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Principal Investigator, William Apro, Ph.D., University of Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_16-200
Record Dates: First submitted 2017-01-19; First posted 2017-01-26 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Amino Acids, Essential

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resting leg of young males (Experimental)
  Interventions: Dietary Supplement: Essential amino acids
- Exercising leg of young males (Experimental)
  Interventions: Dietary Supplement: Essential amino acids
- Resting leg of elderly males (Experimental)
  Interventions: Dietary Supplement: Essential amino acids
- Exercising leg of elderly males (Experimental)
  Interventions: Dietary Supplement: Essential amino acids

INTERVENTIONS:
Dietary Supplement: Essential amino acids — 240 mg essential amino acids per kg body weight dissolved in 500 ml of water provided after exercise.

SUMMARY:
Age-associated loss of muscle mass, termed sarcopenia, is strongly associated with functional impairment and physical disability in the elderly. Maintenance or growth of muscle mass is mainly driven by increased muscle protein synthesis (i.e. the generation of new muscle protein) in response to exercise and feeding. However, several investigations have shown that elderly individuals have a blunted protein synthetic response following protein intake. This inability of the elderly to properly respond to growth stimuli has been termed anabolic resistance and plays a significant role in the development of sarcopenia. However, the precise mechanisms underpinning anabolic resistance are unknown.

It is well established that muscle protein synthesis at the molecular level is regulated by a cellular protein complex called mTORC1. When exposed to a growth stimulus, mTORC1 has been shown to associate with lysosomes, i.e. the intracellular organelles responsible for the breakdown of cellular proteins, and subsequently moving towards the cell periphery.

This movement of lysosome-associated mTORC1 within the cell is believed to be vital for the activation of protein synthesis, as inhibition of lysosomal movement blunts mTORC1 activation in response to amino acids. Thus, dysregulation of lysosomal movement in ageing muscle may represent an underlying mechanism in the development of anabolic resistance. However, this area of research is unexplored in the context of human skeletal muscle. The investigators hypothesize that dysregulation of lysosomal movement plays a central role in the development of age-associated skeletal muscle anabolic resistance.

ELIGIBILITY:
Inclusion Criteria:

Be a non-smoking male within the specified age range for each group (young; 18-35 yrs, old; 65-75 yrs)

Have a BMI (body mass index, body weight/height in m2) between 18 and 25 kg/m2, which is considered a normal body mass index.

Be in good general health: no cardiovascular diseases or metabolic diseases.

Exclusion Criteria:

Health problems such as: heart disease , metabolic disease such as phenylketonuria, rheumatoid arthritis, uncontrolled hypertension, poor lung function, or any health condition that might put the participant at risk when participating in this study.

Generalized neuromuscular disease (such as Parkinson's disease or motorneuron disease).

Involvement in regular structured resistance exercise training at the time of the study.

Consumption of any analgesic drugs, anti-inflammatory drugs, or medication that is known to affect protein metabolism (beta-blockers, corticosteroids, NSAIDs).

Participants who have undergone muscle biopsy testing or isotope infusion procedures within the last 5 years.

Allergic to lidocaine

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-08-30 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
Lysosomal movement | ~360 minutes
  Changes in intracellular localization of lysosomes will be measured via immunofluorescence

SECONDARY OUTCOMES:
Lysosomal movement in isolated muscle cells | ~30 minutes
  Changes in intracellular localization of lysosomes will be measured via immunofluorescence

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport, Exercise and Rehabilitation Sciences at University of Birmingham, Birmingham, West Midlands, United Kingdom